CLINICAL TRIAL: NCT07070726
Title: UNderstanding The Experience of Ovarian Cancer Life After Diagnosis (UNTOLD) Study
Brief Title: UNTOLD Ovarian Cancer Unmet Needs Survey
Status: Recruiting | Type: Observational
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2024LS181; 1U48DP006876 (NIH)
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; quality of life; cancer survivorship
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ovarian Cancer Survivors: Ovarian cancer survivors participate in UNTOLD by completing a one-time survey regarding their experiences

SUMMARY:
The goal of this study is to comprehensively measure ongoing concerns and unmet needs of individuals living with ovarian cancer. To accomplish this, the UNderstanding The experience of Ovarian cancer - Life after Diagnosis (UNTOLD) study will be conducted using a mixed-methods approach. Ovarian cancer survivors will be enrolled to participate in UNTOLD to complete a one-time survey regarding their experiences. Up to 40 survivors will be subsequently identified to complete a follow-up interview. To ensure these sample sizes, along with a representative sample, a combined recruitment strategy will be employed using the California Cancer Registry (population-based) and recruitment through ovarian cancer advocacy groups.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and write in English
* Diagnosed with ovarian cancer (ovarian, primary peritoneal, fallopian tube)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ovarian cancer survivors will be enrolled to participate in UNTOLD to complete a one-time survey regarding their experiences.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Supportive Care Needs | Day 1
  Composite Supportive Care Needs Survey - Short Form (SCNS-SF34) score minimum: 34, maximum: 170; continuous score; presented as mean and standard deviation.

SECONDARY OUTCOMES:
Quality of Life - Average FACT general total score | Day 1
  FACT-General total score minimum 0, maximum 108; continuous score; presented as mean and standard deviation

CONTACTS AND LOCATIONS:
Locations (1):
- Masonic Cancer Center, Minneapolis, Minnesota, United States